CLINICAL TRIAL: NCT01444976
Title: The Effect of Sedation During Transesophageal Echocardiography on Heart Rate Variability:A Comparison of Hypnotic Sedation With Medical Sedation
Brief Title: The Effect of Sedation During Transesophageal Echocardiography on Heart Rate Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Gonenc, Cardiology Clinic, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yuksel-dogan-2011
Record Dates: First submitted 2011-05-26; First posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Transesophageal Echocardiography
Keywords: age range of 18-83
MeSH Terms: interventions — Anesthesia, Local; Hypnosis; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- topical pharyngeal anesthesia (Active Comparator): There were 26 patients who had the procedure under topical pharyngeal anesthesia.
  Interventions: Drug: local anesthesia; Behavioral: hypnosis
- midazolam (Active Comparator): There were 25 patients who received midazolam.
  Interventions: Behavioral: hypnosis; Drug: Midazolam
- hypnosis (No Intervention): There were 27 patients receiving hypnosis.

INTERVENTIONS:
Drug: local anesthesia — patients will receive only topical anesthesia with 1% lidocaine
  Arms: topical pharyngeal anesthesia
Behavioral: hypnosis — Hypnosis will be performed by the same anesthesiologist according to indirect Erickson's method
  Arms: midazolam; topical pharyngeal anesthesia
Drug: Midazolam — Before insertion of the probe, the patients will be sedated with midazolam at a dose of 0,.05 mg/kg iv (to achieve a Ramsay Sedation Score of 2-3). If needed, additional iv doses (0.005 mg/kg) were given during the procedure.
  Arms: midazolam

SUMMARY:
There is no ideal sedation technique that can be used during Transesophageal Echocardiography (TEE), and the data concerning the effects of available sedation techniques on Heart Rate Variability (HRV) are limited. In this study the investigators aimed at comparing the effects of sedation through hypnotherapy with medical sedation achieved by midazolam on HRV.

DETAILED DESCRIPTION:
Seventy-six patients with an indication of TEE will be recruited, the age range will be 18-83 years. In Group Topical (T) there are 26 patients who had the procedure under topical pharyngeal anesthesia, in Group Midazolam (D) there are 25 patients who will receive midazolam and in Group H there are 27 patients receiving hypnosis. All patients will have an IV access; throughout the procedure heart rate, rhythm ECG, peripheric O2 saturation will be monitored with a non-invasive monitor, blood pressure measurements were taken every 3 minutes. Rhythm Holter recordings will be obtained from all patients and TEE will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a need of transesophageal echocardiography

Exclusion Criteria:

* Heart failure
* Bad overall condition
* Arrhythmia

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Hypnotic sedation | two months
  Contrary to sedation with midazolam; when hypnosis is used for sedation in TEE patients, autonomic cardiac tone is modified to a significant extent. Hypnotic sedation achieves this by increasing the parasympathetic activity, decreasing the sympathetic activity and changing the sympathovagal interaction balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Bakırköy, Istanbul, Turkey (Türkiye)